CLINICAL TRIAL: NCT02499055
Title: Internet Based Self-help Therapy With FearFighter™ Versus no Intervention for Anxiety Disorders in Adult Persons: a Randomised Feasibility Trial
Brief Title: A Randomised Feasibility Trial With Internet Based Self-help Therapy
Acronym: IBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); TrygFonden, Denmark (Industry); Student Counselling Service, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FearFighter-RHP2015
Record Dates: First submitted 2015-07-01; First posted 2015-07-15 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Anxiety
Keywords: anxiety; behaviour therapy; computer assisted therapy; psychotherapy
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapy, Computer-Assisted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FearFighter (Experimental): The experimental group will use the program FearFighter™.
  Interventions: Behavioral: FearFighter
- Control group (No Intervention): The control group receive no intervention for nine weeks.

INTERVENTIONS:
Behavioral: FearFighter — FearFighter™ is a nine session cognitive behavioural self-help therapy program delivered over the internet during nine weeks. Each session on FearFighter excluding the homework takes about 30-40 minutes to finish. A support person will make a weekly contact of 10 minutes in average to secure understanding of the program and compliance.
  Other Names: Internet based therapy; Computer assisted therapy
  Arms: FearFighter

SUMMARY:
Background. In Denmark, about 350,000 persons suffer from anxiety. Public health-care services plan to implement internet based self-help psychotherapy (IBT) to be an important alternative and supplement to ordinary face-to-face therapy. Meta-analyses indicate that the effect of IBT for anxiety disorders seems better than no intervention, and in some instances equal to 'usual therapy'. But studies have been characterised by small sample sizes, high risk for bias, including high dropout.

Objective. The objective of this pilot trial is to assess the feasibility of conducting a larger confirmatory trial investigating the benefits and harms of an internet-based self-help therapy program, FearFighter™, compared with no intervention for persons with an anxiety disorder.

Design. An investigator-initiated feasibility randomised clinical trial investigating internet-based therapy with FearFighter™ compared with no intervention for persons with an anxiety disorder. We will include 64 participants.

Eligibility criteria. Inclusion criteria: age 18 or older; specific phobia, panic disorder, agoraphobia, or social phobia is the primary diagnosis according to the DSM-IV; and informed consent. Exclusion criteria: suicidal risk; ongoing episode of bipolar disorder or psychosis; concurrent psychological treatment for the anxiety disorder; unable to attend the intervention; or lack of informed consent.

Intervention. The intervention group will use the program FearFighter™, a nine session cognitive behavioural self-help therapy program delivered over the internet during nine weeks. The control group receive no intervention for nine weeks.

Outcomes. Feasibility outcomes are the fraction that are eligible, the fraction that are randomised, and the compliance in the intervention group. Clinical exploratory outcomes are: remission, Beck Anxiety Inventory, Symptom Check List-90R, WHO Well-Being Index, Sheehan Disability Scale, serious adverse events, and behaviour log from FearFighter.

Time schedule. Participants will be included in the trial from July 2015. Results are expected in February 2016.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Specific phobia, panic disorder, agoraphobia or social phobia is the primary diagnosis according to the DSM-IV
* Written informed consent.

Exclusion Criteria:

* Acute suicidal risk.
* Ongoing episode of bipolar disorder or psychosis.
* Receive concurrent psychological treatment for an anxiety disorder
* Considered unable to attend IBT sessions as planned (due to vacation, work/study placement, sickness or similar occurrences).
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Fractions of participants that are eligible and can be randomised | up to week 10
  We will determine the fraction of potential participants as the number of eligible persons compared to the number of randomised persons. Here, we consider eligible participants' to be persons who fulfill the inclusion criteria. Exclusion criteria and informed consent is not included in this definition of eligibility.
Fraction of participants randomised to the experimental group that will comply with the experimental intervention | up to week 10
  We will determine the fraction of participants randomised to the experimental group that will comply with the experimental intervention, defined as completing at least 6 of 9 FearFighter™ sessions during the intervention
Proportion of participants who fulfil the diagnostic criteria for an anxiety disorder at the end of the intervention measured with 'Mini International Neuropsychiatric Interview' (M.I.N.I.) | up to 37 weeks after start of intervention
  Participants are diagnostic assessed with the 'Mini International Neuropsychiatric Interview' (M.I.N.I.), a short structured interview for the most important psychiatric axis 1 diagnoses in DSM-IV and in ICD-10.

SECONDARY OUTCOMES:
Symptoms: Beck Anxiety Inventory (BAI) | Baseline, 10 weeks and 37 weeks after start of intervention
  Beck Anxiety Inventory (BAI) is a 21-items general questionnaire for anxiety symptoms during the last 14 days.
Symptoms: Symptom check list-90R (SCL-90R) | Baseline, 10 weeks and 37 weeks after start of intervention
  Symptom check list-90R (SCL-90R) is a 90-item questionnaire measuring psychological distress and psychopathology (35). Within SCL-90R we use:
  * Global severity index (GSI);
  * Interpersonal sensitivity subscale;
  * Anxiety subscale; and
  * Phobic anxiety subscale.
Functionality: Sheehan Disability Scale (SDS) | Baseline, 10 weeks and 37 weeks after start of intervention
  Sheehan Disability Scale (SDS). We assess:
  * Occupational function;
  * Social function; and
  * Family function.
Quality of life: WHO Well-Being Index | Baseline, 10 weeks and 37 weeks after start of intervention
  WHO Well-Being Index.,We assess the quality of life.
Serious adverse events (SAE) | SAE will be registrered throughout the intervention from week 0 to week 10
  Serious adverse events, defined as any adverse event that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or is a congenital anomaly or birth defect.
  Other adverse events, defined as any undesirable medical event occurring to a participant during a clinical trial, which does not necessarily have a causal relationship with the intervention.

OTHER OUTCOMES:
Behaviour log from FearFighter | Behaviour log will be registrered throughout the intervention from week 0 to week 10
  Registration of the number of times the participant log on FearFighter.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Lau, MD, Study Director — Stolpegaard Psychotherapy Centre. Mental Health Services in the Capital Region of Denmark.
Locations (1):
- Psychotherapy Center Stolpegård, Mental Health Services in the Capital Region of Denmark, Gentofte Municipality, Capital Region, Denmark

REFERENCES:
- [Derived] Fenger M, Lindschou J, Gluud C, Winkel P, Jorgensen L, Dybkjaer JH, Lau M. Internet-based therapy with FearFighter for anxiety disorders: a randomised clinical trial. Nord J Psychiatry. 2020 Oct;74(7):518-524. doi: 10.1080/08039488.2020.1755363. Epub 2020 May 13. PMID 32401099
- [Derived] Fenger M, Lindschou J, Gluud C, Winkel P, Jorgensen L, Kruse-Blinkenberg S, Lau M. Internet-based self-help therapy with FearFighter versus no intervention for anxiety disorders in adults: study protocol for a randomised controlled trial. Trials. 2016 Oct 28;17(1):525. doi: 10.1186/s13063-016-1619-3. PMID 27793181